CLINICAL TRIAL: NCT06888544
Title: Effects of High-Intensity Interval Training on Bone Health, Physical Fitness and Quality of Life in Elderly Women With Osteopenia: A Pilot Randomized Controlled Trial
Brief Title: Effects of High-Intensity Interval Training on Bone Health in Hong Kong Older Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMRF07220048
Record Dates: First submitted 2025-02-04; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-12

CONDITIONS: Osteopenia
Keywords: Osteopenia; Older women; High-intensity interval training
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: The present research follows a randomized controlled experimental design (RCT), parallel type with two groups in multi-centers, and is assessed in a pretest, posttest, and six months after the completion of the intervention. The participants will be randomly allocated to one experimental group, and one non-exercise control group. The non-exercise control group will be asked to attend a workshop. At the same time, the exercise group performs a HIIT program.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (HIIT) (Experimental): HIIT program for 24 weeks with a frequency of 2 times per week.
  Interventions: Behavioral: HIIT program for 24 weeks with a frequency of 2 times per week.
- Non-exercise control (Placebo Comparator): Participants will not receive any exercise training but will attend 48 recreation workshops.
  Interventions: Behavioral: Non-exercise control

INTERVENTIONS:
Behavioral: HIIT program for 24 weeks with a frequency of 2 times per week. — Participants will receive a 24-week HIIT program, with 2 sessions per week. Each session will comprise three sections, including warm-up, main exercise and cool down. The time will be between 37 to 40 minutes with progression of training. Each HIIT section will include six high-impact weight-bearing exercise. For Weeks 1-4, the HIIT section will include 12 intervals of 30 seconds HIIT workout at corresponding intensity, separated by 11 intervals of 60 seconds of active recovery. To ensure the subjects' safety, a chair will be used for assistance during training in the first month. Additionally, a 3 kg weight will be incorporated for the training in the final two months.
  Arms: High-intensity interval training (HIIT)
Behavioral: Non-exercise control — Workshop participants in the non-exercise control group will receive a series of workshops related to daily recreation.
  Arms: Non-exercise control

SUMMARY:
Osteoporosis is an age-related disease, characterized by a decreased bone mass and an increased risk of fragility fractures. Osteoporosis leads to increasing mortality, disabilities, morbidity of chronic pain, and the cost of health and social care, as well as decreasing the quality of life from reduced independence and hindered physical, mental, and social well-being.

A recent review and meta-analysis, investigating the association between physical activity and osteoporosis prevention in elderly people, indicated that the traditional exercise interventions (i.e., resistance training) were undertaken for 60+ mins, 2-3 times/week for 7+ months. However, participation rates remain low in these exercise programs among older adults, in part due to a need for specialized equipment and correct techniques to prevent injury. In addition, low motivation and associated compliance with such conventional exercise is problematic among older adults.

Considering there is little evidence of HIIT benefits related to older women with osteopenia, the current study aims to evaluate the effectiveness of a 24-week HIIT intervention on bone mineral density, bone turnover markers and other health-related outcomes among Hong Kong Chinese older women.

DETAILED DESCRIPTION:
The study will be a randomized controlled trial (RCT) with two groups and three times repeated measures. Data will be collected in a pretest, post-test, and six months after the intervention. The eligible participants will be randomly distributed into one of two groups in a ratio of 1:1. The participants recruited and meeting the screening criteria will receive a 24-week HIIT intervention or recreation workshop. The intervention effects will be evaluated on bone mineral density, bone turnover markers, physical fitness, fear of falling, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* • 60 to 74 years at the start date of the project

  * diagnosed with osteopenia by DXA scan screening with a BMD at the femoral neck or total hip or lumbar spine between -1 and -2.5 SD T-score below the average values
  * Passing the PAR-Q plus screening or with the physician's approval for readiness to participate in high-intensity exercise
  * Above the average level of 2-mins stepping showing competent aerobic fitness
  * No restriction on physical mobility
  * No cognitive impairment, as determined by the Chinese version of the Mini-Mental Status Examination (i.e., score < 24)
  * No previous substantial experiences in practicing HIIT. The written informed consent form will be collected from each participant

Exclusion Criteria:

* • Severe chronic disease restricting high-intensity exercise

  * Having cognition impairment regarded by specialists
  * checked through medical records at HA Go app platform in the past 6 months, have concurrent medical conditions (e.g., thyrotoxicosis or hyperparathyroidism, Paget's disease, renal disease, diabetes, knee or hip osteoarthritis) and use medications (e.g., corticosteroids, estrogen, thyroxine, thiazide diuretics, or antiretroviral agents) known to affect bone metabolism during past 2 years
  * any condition with osteoporosis, osteoporotic fractures
  * current smoker
  * alcohol 3 or more units per day.

Ages: 60 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 24-weeks intervention (T2 post-test), and 6 months after intervention completion (T3 follow-up test).
  Bone mineral density at the non-dominant lumbar spine and femoral neck of hip will be measured by one registered technician using DXA (XR-46, Norland, Wisconsin, USA) at an assessment center in the Chinese University of Hong Kong.
Bone turnover markers | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 24-weeks intervention (T2 post-test), and 6 months after intervention completion (T3 follow-up test).
  The two bone turnover markers, P1NP (ng/ml) and CTX (ng/L) will be used to assess the subjects' bone formation and bone resorption. Participants must arrive at the elderly center between 08:30 and 09:30 a.m. after a 12-hour overnight fast and avoid intense physical activity the night before. A qualified nurse will collect 5 mL of venous blood from the antecubital vein, which will coagulate at room temperature for 20-30 minutes before being transported to the lab within one hour. The blood will then be centrifuged at 4 °C and 3000 rpm for 50 minutes, with the resulting sample stored at -80 °C for serum biochemical marker assays. Serum P1NP and CTX levels will be measured using ELISA kits from Immunodiagnostic Systems Inc., and analysis will be conducted by the Hong Kong Polytechnic University test lab.

SECONDARY OUTCOMES:
Physical fitness_Body mass index | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 24-weeks intervention (T2 post-test), and 6 months after intervention completion (T3 follow-up test).
  BMI (kg/m²) was calculated by dividing weight in kilograms by the square of height in meters. Body weight was measured using a mobile scale that was accurate to 0.01 kg and calibrated before use. Participants were instructed to remain still until the digital display stabilized, at which point their weights were recorded. Height was measured using a mobile stadiometer accurate to 0.1 cm, and participants were asked to stand straight with their knees together during the measurement.
Physical fitness_Lower limb muscle strength | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 24-weeks intervention (T2 post-test), and 6 months after intervention completion (T3 follow-up test).
  30-Second Chair Stand will used to assess lower limb muscle strength. The required tools will include a straight-backed chair (43 cm seat height) and a timer. Participants will sit in the middle of the chair with their feet shoulder-width apart, crossing their arms at the wrists close to their chest. They will then stand fully and sit back down, counting this as one movement, which will be repeated for 30 seconds after the initial instruction.
Physcal fitness_Upper limb muscle strength | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 24-weeks intervention (T2 post-test), and 6 months after intervention completion (T3 follow-up test)
  30-second Arm Curl will be used to evaluate upper limb muscle strength. This test will measure upper body strength using a 5-pound dumbbell, a chair without armrests, and a timer. Conducted on the stronger arm, participants will curl their arm through a full range of motion, turning the palm upward. They will fully bend and straighten the arm at the elbow, repeating this as many times as possible within 30 seconds.
Physical fitness_Aerobic endurance | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 24-weeks intervention (T2 post-test), and 6 months after intervention completion (T3 follow-up test).
  Aerobic endurance will be measured by a 2-Minute Step Test. A timer will be used for this procedure. Participants will stand straight next to a wall, where a mark will indicate the midpoint between the kneecap and hip bone. They will step for two minutes, lifting their knees to the mark's height.
Physical fitness_Lower body flexibility | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 24-weeks intervention (T2 post-test), and 6 months after intervention completion (T3 follow-up test).
  Lower body flexibility will be assessed by a Chair Sit-and-Reach Test. The required tools will include a ruler and a straight-backed chair about 43 cm high. Participants will sit on the edge of the chair, with one foot flat on the floor and the other leg extended forward, keeping the knee straight and the ankle at a 90° angle. They will reach forward toward their toes with overlapping hands, maintaining a straight back and keeping their heads up. The distance from their fingertips to their toes will be measured and held for a moment.
Physical fitness_Upper body flexibility | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 24-weeks intervention (T2 post-test), and 6 months after intervention completion (T3 follow-up test).
  Upper body flexibility will be assessed by the Back Scratch Test. The required tool will be a ruler. Participants will place one hand behind their head and over their shoulder, reaching as far as possible with the palm against the body and fingers pointing down. The other arm will be positioned behind the back, with the palm facing outward and fingers pointing up, reaching to overlap the fingertips of both hands. The distance between the tips of the middle fingers will be measured.
Physical fitness_Mobility and dynamic balance | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 24-weeks intervention (T2 post-test), and 6 months after intervention completion (T3 follow-up test).
  Mobility and dynamic balance will be measured by the 8-Foot Up-and-Go Test. The required tools will include a timer, a straight-backed chair about 43 cm high, a cone marker, and a measuring tape. The cone will be placed 2.4 m in front of the chair. Participants will start by sitting with their hands on their knees and feet flat on the ground. They will then stand up and walk quickly (without running) to round the cone and return to sit down. The time taken from standing to sitting will be measured.
Fear of falling | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 24-weeks intervention (T2 post-test), and 6 months after intervention completion (T3 follow-up test).
  Fear of falling (FOF) will be measured using the Chinese version of the Falls Efficacy Scale-International (FES-I). This scale includes questions adapted from the original 16-item FES-I questionnaire to evaluate FOF during specific daily activities. The total score of the questionnaire ranges from 16 to 64, and a higher score indicates that the individual perceives themselves as having a significant fear of falling, which can lead to reduced activity levels and an increased risk of social isolation. The Chinese version of SFES-I demonstrated good internal consistency and reliability, with a Cronbach's α of 0.88.
Perceived quality of life | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 24-weeks intervention (T2 post-test), and 6 months after intervention completion (T3 follow-up test).
  The quality of life will be assessed using the brief version of the Hong Kong Chinese WHO Quality of Life Scale (WHOQOL-BREF) (Cronbach's α = .73 - .84). The scale includes 28 items, covering four dimensions of how older adults perceive their quality of life. The total score of the questionnaire ranges from 28 to 140, and a higher score indicates that the individual feels they have a high quality of life.

OTHER OUTCOMES:
Heart rate | Heart rate will be monitored from the start of warm-up to the end of cool-down at each exercise session during the 24-weeks exercise intervention.
  Participants will be monitored by Polar verity sensor during exercise and their heart rate will be monitored to ensure their safety and intensity adherence of exercise protocol.
Self-reported Rate of Perceived Exertion (RPE) | RPE will be asked at the end of main exercise at each exercise session during the 24-weeks intervention
  Older women will be asked about the self-reported Rate of Perceived Exertion (RPE Borg CR-10 category scale) after they complete the main exercise training in each session. A higher score (closer to 10) means the individual feels they are working much harder, while a lower score (closer to 0) suggests a much easier level of activity.
Safety: adverse events | Adverse events will be asked at the end of each exercise session during the 24-weeks intervention program
  All adverse events will be recorded as safety endpoints.
Exercise acceptability | The exercise acceptability will be evaluated after 24 weeks of intervention.
  Exercise acceptability will be assessed post-intervention using ten questionnaire items responding to a 5-point Likert scale (strongly disagree, disagree, neither agree nor disagree, agree, and strongly agree). The score on this scale ranges from 9 to 40, the higher score shows better acceptability to the exercise intervention.
Process evaluation of intervention program | Outcome evaluations will be conducted at the completion of 24-weeks intervention
  A process evaluation scale of the intervention process will be developed for this study based on the previous framework of process evaluation for the intervention study. This scale with 10 items using a 5-point (strongly unsatisfied, unsatisfied, neutral, satisfied, and strongly satisfied). The score on this scale ranges from 10 to 50, a higher score shows higher satisfaction with the intervention program.
Retention rate | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 24-weeks intervention (T2 post-test), and 6 months after intervention completion (T3 follow-up test).
  Percentage of participants completing assessments at the pre-intervention test, post-intervention test and follow up test
Session attendance rate | Session attendance will be recorded during the 24-week intervention
  Percentage of participants completed at least 75% of intervention sessions (36/48 sessions).

CONTACTS AND LOCATIONS:
Overall Officials: Yanping Duan, Principal Investigator — Hong Kong Baptist University; Department of Sport, Physical Education and Health
Locations (1):
- Bliss District Elderly Community Centre, China, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chapman, J. J., Coombes, J. S., Brown, W. J., Khan, A., Chamoli, S., Pachana, N. A., & Burton, N. W. (2017). The feasibility and acceptability of high-intensity interval training for adults with mental illness: A pilot study. Mental Health and Physical Activity, 13, 40-48
- [Background] Grant A, Treweek S, Dreischulte T, Foy R, Guthrie B. Process evaluations for cluster-randomised trials of complex interventions: a proposed framework for design and reporting. Trials. 2013 Jan 12;14:15. doi: 10.1186/1745-6215-14-15. PMID 23311722
- [Background] Kwan MM, Tsang WW, Close JC, Lord SR. Development and validation of a Chinese version of the Falls Efficacy Scale International. Arch Gerontol Geriatr. 2013 Jan-Feb;56(1):169-74. doi: 10.1016/j.archger.2012.10.007. Epub 2012 Oct 30. PMID 23116978
- [Background] Marriott CFS, Petrella AFM, Marriott ECS, Boa Sorte Silva NC, Petrella RJ. High-Intensity Interval Training in Older Adults: a Scoping Review. Sports Med Open. 2021 Jul 19;7(1):49. doi: 10.1186/s40798-021-00344-4. PMID 34279765
- [Background] Carlson SA, Fulton JE, Schoenborn CA, Loustalot F. Trend and prevalence estimates based on the 2008 Physical Activity Guidelines for Americans. Am J Prev Med. 2010 Oct;39(4):305-13. doi: 10.1016/j.amepre.2010.06.006. PMID 20837280
- [Background] Zitzmann AL, Shojaa M, Kast S, Kohl M, von Stengel S, Borucki D, Gosch M, Jakob F, Kerschan-Schindl K, Kladny B, Lange U, Middeldorf S, Peters S, Schoene D, Sieber C, Thomasius F, Uder M, Kemmler W. The effect of different training frequency on bone mineral density in older adults. A comparative systematic review and meta-analysis. Bone. 2022 Jan;154:116230. doi: 10.1016/j.bone.2021.116230. Epub 2021 Oct 5. PMID 34624560
- [Background] Lin CY, Park JH, Hsueh MC, Sun WJ, Liao Y. Prevalence of Total Physical Activity, Muscle-Strengthening Activities, and Excessive TV Viewing among Older Adults; and Their Association with Sociodemographic Factors. Int J Environ Res Public Health. 2018 Nov 8;15(11):2499. doi: 10.3390/ijerph15112499. PMID 30413089
- [Background] Pinheiro MB, Oliveira J, Bauman A, Fairhall N, Kwok W, Sherrington C. Evidence on physical activity and osteoporosis prevention for people aged 65+ years: a systematic review to inform the WHO guidelines on physical activity and sedentary behaviour. Int J Behav Nutr Phys Act. 2020 Nov 26;17(1):150. doi: 10.1186/s12966-020-01040-4. PMID 33239014
- [Background] Nguyen VH. Osteoporosis prevention and osteoporosis exercise in community-based public health programs. Osteoporos Sarcopenia. 2017 Mar;3(1):18-31. doi: 10.1016/j.afos.2016.11.004. Epub 2016 Dec 24. PMID 30775499